CLINICAL TRIAL: NCT06678672
Title: Contingency Management for Veteran Smokers Undergoing Major Elective Surgery
Acronym: CM_Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Tobacco Related Disease Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-41632
Record Dates: First submitted 2024-11-04; First posted 2024-11-07 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Tobacco Use Disorder; Substance Use Disorder (SUD)
Keywords: Tobacco; Contingency Management; Surgery
MeSH Terms: conditions — Tobacco Use Disorder; Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This is a pilot randomized-controlled trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contingency Management (CM) (Experimental): A VA CM Protocol will be established after gathering feedbacks from focus groups with Veterans and advice from the experts in 1) surgical care, 2) CM, and 3) VA policy. The CM intervention group will follow the established VA CM Protocol to deliver treatment over 5 weeks. The participants in the CM group will also be offered a 5-week supply of medication for Tobacco Use Disorder (TUD).
  Interventions: Behavioral: Contingency Management (CM)
- Treatment as Usual (TAU) (Active Comparator): Participants assigned to TAU will receive usual care at San Francisco VA Health Care System (referral to Tobacco Cessation Clinic and the VA Telequit Quitline) over the 5 weeks. They will also be offered a 5-week supply of medication for Tobacco Use Disorder (TUD).
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Contingency Management (CM) — The participants will receive and be trained to use a CO monitor and iCO app to upload videos to verify smoking abstinence at a minimum of once per day, 5 times per week, over 5 weeks. Financial incentives will be provided at weekly visits contingent on tobacco abstinence verified through remote CO monitoring. They will receive clinician feedback at the time of each CO reading, following the established VA CM protocol developed in the earlier phase of the project. Each CO reading during the weeks 2-5 will also be accompanied with a brief (5-minute) telephone or video feedback CM counseling session from the study clinician.
  Arms: Contingency Management (CM)
Behavioral: Treatment as Usual (TAU) — Participants assigned to TAU will receive usual care at San Francisco VA Health Care System (SFVAHCS), i.e., referral to Tobacco Cessation Clinic and the VA Telequit Quitline. The SFVAHCS Tobacco Cessation Clinic is a consult service that calls patients proactively 3 times to offer 1:1 behavioral counseling for smoking cessation. VA Telequit is a national toll-free number available to Veterans that allows them to speak with a smoking cessation counselor for up to 5 sessions per NCI Quitline guidelines. The smoker initiates the first call, and subsequent calls will be proactively made by Quitline staff.
  Arms: Treatment as Usual (TAU)

SUMMARY:
The goal of this study is to design and test the first mobile contingency management (CM) smoking cessation intervention for military Veterans undergoing major elective surgery. Smoking is the leading risk factor for postoperative complications and is associated with longer hospital stays, reoperations, and 30-day mortality. Smoking rates among patients undergoing major elective surgery are high, 22.3-43.0%. It is imperative to identify efficacious, strategically timed smoking cessation interventions for surgery patients.

CM incentivizes smoking cessation through positive reinforcement (rewards) when bioverified abstinence is achieved. To ensure feasibility, CM must be tailored to the clinical context. CM for smoking cessation has never been delivered before and after major surgery, nor has mobile CM bioverification been trialed perioperatively. The investigators will develop and test a tailored mobile smoking cessation CM protocol for Veterans undergoing major elective surgery.

DETAILED DESCRIPTION:
Major elective surgery is common among Veterans and smoking is the most significant modifiable risk factor for perioperative morbidity and mortality. Major elective surgeries, including general, thoracic, vascular, urologic, spinal, orthopedic, and other surgeries, are common in the Veterans Affairs (VA) Healthcare System, with over 600,000 surgical procedures occurring annually across the VA. Reducing complications and death after major elective surgery is a top priority, both for Veterans and the general population. Smoking at the time of surgery is the single greatest risk factor for complications, reoperation, and death. The relative risk (RR) of death is 1.53 times higher in the 30 days after major surgery in smokers compared to non-smokers. Smoking before all types of surgeries is associated with postoperative pneumonia, prolonged intubation, myocardial infarction, stroke; infections, sepsis, and poor wound healing; and repeat procedures. Smoking at the time of surgery has additive risk of postoperative mortality when patients have other modifiable risk factors such as poor nutritional status, hyperglycemia, and alcohol use.

Contingency management (CM) is an efficacious, scalable behavioral intervention for smoking cessation in patients with tobacco use disorder (TUD). CM is a behavioral treatment that uses positive reinforcement to incentivize behavior change by delivering financial rewards (i.e., vouchers, cash equivalent) when the target behavior is achieved and biologically verified. It is feasible for Veterans with substance use disorder (SUD) and has been implemented widely across the VA. However, the CM protocol still needs to be tested out and evaluated to tailor for the clinical population.

The investigators will develop and test a tailored mobile smoking cessation contingency management (CM) protocol for Veterans undergoing major elective surgery. First, the investigators will adapt a CM protocol for delivery over 5 weeks using mobile CO monitoring in the perioperative period. To ensure acceptability, the investigators will consult with a Community Advisory Panel (CAP) of Veteran patient advocates; CM and surgery content experts; and VA policymakers on CM methods, timing, and delivery. The investigators will then conduct a pilot randomized-controlled trial (RCT) in which 36 Veteran smokers undergoing major elective surgery (general, spinal, thoracic, vascular, urological, gynecological, orthopedic, or gender-affirming) will be randomized to receive the 5-week perioperative mobile CM (n=18) or 5-week of treatment as usual (TAU, VA Tobacco Cessation Clinic and Quitline) (n=18). Participants in both conditions will receive pharmacotherapy. This study will demonstrate proof-of-principle of CM delivery perioperatively.

The aims of the study are as follows:

Aim 1: To develop a mobile CM smoking cessation protocol to be integrated into VA surgical settings.

Aim 2: To assess the feasibility of smoking cessation CM for VA surgery patients, measured by 1) Recruitment (ability to recruit ≥70% of the sample), 2) Engagement (≥50% of CM participants completing ≥25% of CM sessions and ≥25% of CO video uploads), and 3) Retention (measure completion in ≥60% of all participants at Week 5 (Study End)).

Aim 3: To compare CM with TAU on improving smoking cessation outcomes (quit attempts, cigarettes per day, and nicotine dependence severity) at Study End (Week 5).

Exploratory Aim: To measure cigarette abstinence in both conditions.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking;
* Veteran enrolled in healthcare at SFVAHCS;
* Veteran scheduled for major elective surgery within the next 6 months (including but not limited to: general, spinal, thoracic, vascular, urological, gynecological, orthopedic, gender affirming). Veterans, who are followed at SFVAHCS by Primary Care and are referred to outside institutions for major surgery (e.g., gynecological or gender-affirming surgeries) are also eligible to participate;
* Current (past 30 days) cigarette smoking a minimum of 1 cigarette per day (average), assessed by Timeline Followback (TLFB);
* Open to receiving smoking cessation interventions.

Exclusion Criteria:

Evaluated by investigative team medical record review and clinical assessment: - Psychotic disorders, bipolar disorder, neurocognitive disorder, or other psychiatric or medical conditions judged by the PI to be unstable based on medical record review and/or screening results;

* Untreated, current, active problem gambling, assessed by medical record diagnosis and/ or Problem Gambling Severity Index (PGSI) score ≥ 8;
* Enrollment in end of life/ palliative care;
* Surgery with a clinical indication for cancer;
* Unable to meet time commitment;
* Currently pregnant or planning to become pregnant during the study (people of childbearing potential ages 18-55);
* A suicide attempt or suicidal ideation with intent in the 30 days before enrollment;
* Concurrent participation in another tobacco cessation trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Recruitment | Up to approximately 20 months
  Ability to recruit ≥70% of the target sample within the study timeline, i.e., at least 25 of 36 participants are enrolled.
Feasibility - Engagement | Weeks 2-5
  It will be measured by the cutting points of ≥50% of participants attending ≥25% CM sessions and ≥25% CO video uploads during Weeks 2-5 in the CM intervention group.
Feasibility - Retention | Weeks 0-5 (Baseline - Week 5)
  It will be measured by a cutting point of ≥60% of enrolled participants completing self-report measures, staff measures, and bioverification over 5 weeks of the study.
Frequency of quit attempts | Weeks 0 - 6 (Baseline - Follow-up)
  Quite attempts (a period of intentionally not smoking for ≥ 24 hours) will be assessed by self-report (Nicotine and Tobacco Use Survey) and confirmed with Timeline Follow-Back (TLFB, past 30 days). Nicotine and Tobacco Use Survey was developed by our team and it will assess age at first use, duration of use, use of all forms of nicotine and tobacco, prior quit attempts (defined as a period of intentionally not smoking for ≥ 24 hours), duration of cessation (if any), and presence of other tobacco users in the home. At Week 5, the survey will also inquire about the frequency and duration of quit attempts in the past 30 days. TLFB uses a calendar with specific anchor dates to identify the quantity and frequency of use.
Amount of Cigarettes per day | Weeks 0 -6 (Baseline - Follow-up)
  Self-report of tobacco use will be assessed by Timeline Followback (TLFB, past 30 days at baseline), which uses a calendar with specific anchor dates to identify the quantity and frequency of use.
Nicotine dependence severity | Weeks 0 & 6 (Baseline & Follow-up)
  Nicotine dependence severity will be assessed through Fagerstrom Nicotine Dependence (FTND). It contains six items that evaluate the quantity of cigarette consumption, the compulsion to use, and dependence. In scoring the Fagerstrom Test for Nicotine Dependence, yes/no items are scored from 0 to 1 and multiple-choice items are scored from 0 to 3. The items are summed to yield a total score of 0-10. The higher the total Fagerstrom score, the more severe the patient's nicotine dependence is.

SECONDARY OUTCOMES:
Cigarette Abstinence | Weeks 1-6 (Week 1 to Follow-up)
  A 7-day point prevalence cigarette abstinence will be defined as 1) no smoking 7 days prior (via TLFB), and 2) CO levels < 6 ppm. For individuals with CO levels > 6 ppm, who report smoking cannabis on TLFB and not receiving Nicotine Replacement Therapy (NRT), salivary cotinine <10 nanograms/ milliliter (ng/ml) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Herbst, MD, Principal Investigator — San Francisco VA Health Care System
Locations (1):
- San Francisco VA Health Care System, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No